CLINICAL TRIAL: NCT05600543
Title: Evaluation of the Effect of Lumbar Belt on Spinal Mobility in Subjects With and Without Low Back Pain
Acronym: LombaMob
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thuasne (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-A01060-43; ANSM (Other: 2022-A01060-43)
Record Dates: First submitted 2022-10-21; First posted 2022-10-31 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2024-09

CONDITIONS: Low Back Pain
Keywords: Low Back Pain; Lumbar belt; Movement; Kinematics
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1: Lumbar belt Lombastab® (Thuasne, Levallois Perret, France) (Experimental): Low back pain patients wear Lumbar belt Lombastab® during 4 weeks according to the instructions given by the investigator of the study.
  Interventions: Device: Lumbar belt
- Optional arm: Healthy subjects who will done the third additional visit (Experimental): For the healthy subjects, they will be offered to do a third additional visit during which they will be able to test the Lombaskin lumbar belt and the Lyne Up percko postural T-shirt.

INTERVENTIONS:
Device: Lumbar belt — All subjects (LBP group and healthy group) wear the belt during the two visits to perform differents tests.
  The invistigator will ask the LBP patients to wear the lumbar belt between the two visits (for 4 weeks, for 4 to 8 hours per day)
  Arms: Arm 1: Lumbar belt Lombastab® (Thuasne, Levallois Perret, France)
Device: Lombaskin lumbar belt and the Lyne Up percko postural T-shirt. — Lombaskin lumbar belt and the Lyne Up percko postural T-shirt could be worn during the third addtional visit proposed to the healthy subject.

SUMMARY:
Low back pain (LBP) is a common condition worldwide as the lifetime prevalence is up to 80%. It is defined as pain in the lumbosacral region in which the etiological causes are most often mechanical, and it is therefore defined as "non-specific LBP".

Lumbar belts are used in the treatment and secondary prevention of LBP. They are supposed to reduce the intensity of pain by improving the functional capacities of daily activities and thus preventing the risk of chronicity related to immobility (HAS).

Despite some proof of their efficiency in the literature, it is still not clear how the pressure applied by the belt and the immobilization constraints on the trunk improve the patient mobility.

Considering that LBP causes movement limitation, and that the lumbar belt contributes to initially decrease the pain intensity, as well as to improve the mobility and the functional capacities of the patient, we propose to evaluate the clinical and biomechanical effects of the lumbar belt during different trunk movements in subjects with and without LBP.

This is a clinical investigation on a CE marked medical device, used in accordance with its intended purpose, in the context of a post-marketing clinical follow-up with additional non-invasive procedures (IC SCAC: case 4.1 of the medical device regulation 2017/745).This is a prospective, monocentric, comparative and open clinical investigation.

The objective is to evaluate the clinical and functional effects related to spinal movements in 2 conditions, with and without the wearing of a lumbar belt. The study will be carried out with two groups of subjects: one group of subjects presenting an episode of LBP (NS>4) (subjects considered to have subacute or chronic nonspecific LBP according to the classification of LBP) and another group of control subjects with no spinal symptoms and no pain that could limit movement (healthy subjects).

Each group will undergo 2 visits on 2 separate days with a 30-day delay for the LBP subjects and a 7-day delay for the healthy subjects

* a first visit (V1) for inclusion, familiarization with a clinical and functional test, and an external measurement of spinal mobility during movements;
* a second visit (V2) for a clinical and functional evaluation, external measurements of spinal mobility and biomechanical measurements.

A third visit (V3) will be offered to healthy subjects for the measurement of spinal segment kinematics with the LombaSkin belt and Percko postural T-shirt.

ELIGIBILITY:
Inclusion Criteria for subjects Low Back Pain:

* Male or female,
* Aged between 18 and 70 years,
* With a waist circumference between 75 cm and 110 cm,
* With a 18.5 < BMI < 30 kg/m2,
* Suffering from a current episode of non-specific low back pain (symptomatic subjects),
* At least one average low back pain at rest or during exercise in the last 72 hours collected at inclusion (≥ 4/10 on an EN scale),
* Followed by a primary care physician or specialist for this clinical condition,
* Having received or scheduled to receive an EOS type radiological workup in less than 6 months
* Affiliated or entitled to a social security system,
* Having signed the written consent.

Inclusion Criteria for healthy subjects:

* Male or female,
* Aged 18 to 70 years,
* With a waist circumference between 75 cm and 110 cm,
* With a 18.5 < BMI < 30 kg/m2,
* Never having suffered from LBP or any other type of lumbar disorder,
* Affiliated or entitled to a social security system,
* Having signed the written consent.

Exclusion Criteria:

* Subjects suffering from LBP of inflammatory, tumoral or infectious cause.
* Pregnant women.
* Subjects with cognitive or mental disorders or confirmed depression;
* Subjects who received an infiltration less than one month prior to the inclusion visit or planned during the study;
* Subjects with a known allergy to any of the materials;
* Subjects complaining of chronic, unstabilized or symptomatic cardiac or respiratory problems;
* Subjects with current participation in an interventional investigational drug or device therapy study that impacts the endpoints.
* Subjects under legal protection or unable to express their consent;
* Subject presenting a lumbar radicular syndrome (hiatal hernia, spinal stenosis...).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2022-09-30 (Actual); Primary Completion 2024-03-29 (Actual); Study Completion 2024-03-29 (Actual)

PRIMARY OUTCOMES:
Spinal Mobility assessed by the fingertip to floor distance test (FTF) | Immediately with and without wearing the lumbar belt (Day 0)
  The effect of wearing a lumbar belt on spinal mobility during anterior flexion of the trunk (sagittal plane) in subjects with LBP using the fingertip to floor (FTF) distance test.
Spinal Mobility assessed by the fingertip to floor distance test (FTF) | After 4 weeks with and without wearing the lumbar belt (Day 30)
  The effect of wearing a lumbar belt (for 4 weeks) on spinal mobility during anterior flexion of the trunk (sagittal plane) in subjects with LBP using the fingertip to floor (FTF) distance test.

SECONDARY OUTCOMES:
Spinal Mobility assessed by the fingertip to floor distance test (FTF) | During the Day 0 (for both groups) and Day 30 (for LBP patients) with and without wearing the belt
  Spinal mobility (using the FTF test in forward flexion, the FTF test in lateral flexion and the sternum to wall test in extension):
  a.1) In subjects with LBP at Day 0 and Day 30
  a.2) In healthy subjects (at Day 0)
  a.3) Between healthy subjects and LBP subjects (at Day 0)
Pain level assessed by Numerical Scale (NS) | During the Day 0 and Day 30 immediately before and after wearing the belt, and after each movement with and without the belt (for LBP patients)
  Pain in LBP subjects (Day 0 vs Day 30) using Numerical Scale (NS) from 0 to 10 (0: no pain and 10: worst pain)
Functional capacities assessed by Oswestry Disability Index (ODI) | During the beginning of Day 0 and Day 30 (for LBP patients)
  Functional capacities of LBP subjects (Day 0 and Day 30) using Oswestry Disability Index (ODI)
Kinematics of the spinal segments assessed by Inertial Measurement Units sensors | During Day 0 (for both groups), third visit (for healthy subjects) and Day 30 (for LBP patients) with and without wearing the belt
  Kinematics of the spinal segments using 3 IMUs (Inertial Measurement Units) sensors:
  d.1) In LBP subjects (Day 0 vs Day 30) d.2) In healthy subjects (at Day 0 and at the third visit only on LombaSkin belt and Percko postural T-shirt) d.3) Between healthy subjects and LBP subjects (at Day 0)
Trunk posture measured by 8-camera image stereo correlation system | During Day 7 (for healthy subjects) and Day 30 (for LBP patients)
  Trunk posture using 8-camera image stereo-correlation system (Alternative to motion capture) e.1) In subjects with LBP (Day 30) e.2) In healthy subjects (at Day 7) e.3) Between healthy subjects and subjects with LBP (Day 7 vs Day 30)
The pressure applied by the belt on the trunk assessed by piezo-resistive sensors | During Day 7 (for healthy subjects) and Day 30 (for LBP patients)
  The pressure applied by the belt on the trunk using piezo-resistive sensors f.1) In subjects with LBP (Day 30) f.2) In healthy subjects (at Day 7) f.3) Between healthy subjects and LBP subjects (Day 7 vs Day 30)
Deformation of the lumbar belt assessed by 8-camera image stereo-correlation system | During Day 7 (for healthy subjects) and Day 30 (for LBP patients)
  To evaluate, during spinal movements, the deformation of the lumbar belt considered as a mechanism of action using 8-camera image stereo-correlation system:
  g.1) In LBP subjects (Day 30) g.2) In healthy subjects (Day 7) g.3) Between healthy subjects and LBP subjects (Day 7 vs Day 30)

CONTACTS AND LOCATIONS:
Overall Officials: Paul CALMELS, MD PhD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- CHU de St Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Oshikawa T, Kaneoka K, Morimoto Y, Akuzawa H. Comparison of Lumbar Kinematics with a History of Low Back Pain During Baseball Hitting. Int J Sports Med. 2020 Feb;41(2):119-127. doi: 10.1055/a-1014-3041. Epub 2020 Jan 7. PMID 31910447
- [Background] Masharawi Y, Haj A, Weisman A. Lumbar Axial Rotation Kinematics in an Upright Sitting and With Forward Bending Positions in Men With Nonspecific Chronic Low Back Pain. Spine (Phila Pa 1976). 2020 Mar 1;45(5):E244-E251. doi: 10.1097/BRS.0000000000003265. PMID 32032339
- [Background] Christe G, Rochat V, Jolles BM, Favre J. Lumbar and thoracic kinematics during step-up: Comparison of three-dimensional angles between patients with chronic low back pain and asymptomatic individuals. J Orthop Res. 2020 Jun;38(6):1248-1256. doi: 10.1002/jor.24575. Epub 2020 Jan 7. PMID 31879969
- [Background] Marich AV, Hwang CT, Sorensen CJ, van Dillen LR. Examination of the Lumbar Movement Pattern during a Clinical Test and a Functional Activity Test in People with and without Low Back Pain. PM R. 2020 Feb;12(2):140-146. doi: 10.1002/pmrj.12197. Epub 2019 Sep 3. PMID 31140705
- [Background] Haj A, Weisman A, Masharawi Y. Lumbar axial rotation kinematics in men with non-specific chronic low back pain. Clin Biomech (Bristol). 2019 Jan;61:192-198. doi: 10.1016/j.clinbiomech.2018.12.022. Epub 2018 Dec 22. PMID 30594767
- [Background] Hernandez A, Gross K, Gombatto S. Differences in lumbar spine and lower extremity kinematics during a step down functional task in people with and people without low back pain. Clin Biomech (Bristol). 2017 Aug;47:46-52. doi: 10.1016/j.clinbiomech.2017.05.012. Epub 2017 May 27. PMID 28600994
- [Background] Mitchell K, Porter M, Anderson L, Phillips C, Arceo G, Montz B, Levy S, Gombatto SP. Differences in lumbar spine and lower extremity kinematics in people with and without low back pain during a step-up task: a cross-sectional study. BMC Musculoskelet Disord. 2017 Aug 25;18(1):369. doi: 10.1186/s12891-017-1721-z. PMID 28841866
- [Background] Shojaei I, Salt EG, Hooker Q, Van Dillen LR, Bazrgari B. Comparison of lumbo-pelvic kinematics during trunk forward bending and backward return between patients with acute low back pain and asymptomatic controls. Clin Biomech (Bristol). 2017 Jan;41:66-71. doi: 10.1016/j.clinbiomech.2016.12.005. Epub 2016 Dec 10. PMID 27992778
- [Background] Gombatto SP, D'Arpa N, Landerholm S, Mateo C, O'Connor R, Tokunaga J, Tuttle LJ. Differences in kinematics of the lumbar spine and lower extremities between people with and without low back pain during the down phase of a pick up task, an observational study. Musculoskelet Sci Pract. 2017 Apr;28:25-31. doi: 10.1016/j.msksp.2016.12.017. Epub 2017 Jan 5. PMID 28171775
- [Background] Marich AV, Hwang CT, Salsich GB, Lang CE, Van Dillen LR. Consistency of a lumbar movement pattern across functional activities in people with low back pain. Clin Biomech (Bristol). 2017 May;44:45-51. doi: 10.1016/j.clinbiomech.2017.03.004. Epub 2017 Mar 7. PMID 28324797
- [Background] Vaisy M, Gizzi L, Petzke F, Consmuller T, Pfingsten M, Falla D. Measurement of Lumbar Spine Functional Movement in Low Back Pain. Clin J Pain. 2015 Oct;31(10):876-85. doi: 10.1097/AJP.0000000000000190. PMID 25503596
- [Background] Gombatto SP, Brock T, DeLork A, Jones G, Madden E, Rinere C. Lumbar spine kinematics during walking in people with and people without low back pain. Gait Posture. 2015 Oct;42(4):539-44. doi: 10.1016/j.gaitpost.2015.08.010. Epub 2015 Sep 3. PMID 26380913
- [Background] Van Hoof W, Volkaerts K, O'Sullivan K, Verschueren S, Dankaerts W. Comparing lower lumbar kinematics in cyclists with low back pain (flexion pattern) versus asymptomatic controls--field study using a wireless posture monitoring system. Man Ther. 2012 Aug;17(4):312-7. doi: 10.1016/j.math.2012.02.012. Epub 2012 Mar 20. PMID 22436688